CLINICAL TRIAL: NCT03520946
Title: A Phase III Study of RAMucirumab in Combination With TAS102 vs. TAS102 Monotherapy in Chemotherapy Refractory Metastatic Colorectal Cancer Patients
Brief Title: RAMucirumab in Combination Wth TAS102 vs. TAS102 Alone in Chemotherapy Refractory Metastatic Colorectal Cancer Patients
Acronym: RAMTAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Eli Lilly and Company (Industry); Trium Analysis Online GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMTAS; 2017-004162-99 (EudraCT Number)
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; ramucirumab; tas102
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ramucirumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (ramucirumab + TAS102) (Experimental): Patients randomized to arm A will receive ramucirumab 8 mg/kg iv over 60 min on d1+15, q4w and TAS102 35mg/m2 p.o. twice daily (BID) d1-5 and 8-12, q4w until progression or intolerance or completion of 6 cycles.
  Interventions: Drug: Ramucirumab; Drug: TAS 102
- Arm B (TAS102 only) (Active Comparator): Patients randomized to arm B will receive TAS102 35mg/m2 p.o. twice daily (BID) d1-5 and 8-12, q4w until progression, intolerance or completion of 6 cycles.
  Interventions: Drug: TAS 102

INTERVENTIONS:
Drug: Ramucirumab — 8 mg/kg iv over 60 min on d1+15, q4w
  Arms: Arm A (ramucirumab + TAS102)
Drug: TAS 102 — 35mg/m2 p.o. twice daily (BID) d1-5 and d8-12, q4w

SUMMARY:
Interventional, prospective, randomized (1:1), controlled, open label, multicenter phase IIb study in patients with advanced metastatic colorectal cancer. The scope of the trial is to evaluate overall survival of either regimen (TAS102 +/- Ramucirumab) and evaluate safety and tolerability.

DETAILED DESCRIPTION:
This is an interventional, prospective, randomized (1:1), controlled, open label, multicenter phase IIb study in patients with advanced metastatic colorectal cancer. The scope of the trial is to evaluate overall survival of either regimen and evaluate safety and tolerability.

Patients with advanced metastatic and inoperable, colorectal cancer who have progressed on/after or did not tolerate: fluoropyrimidines, oxaliplatin, irinotecan, anti-angiogenic therapies (bevacizumab, aflibercept, regorafenib or ramucirumab) and when indicated anti-EGFR (epidermal growth factor receptor) antibodies (cetuximab or panitumumab) will be included in this trial.

Patients will be stratified by the duration of previous anti-angiogenic therapy ≥ or <12 months in total, BRAF V600E mutation status (mutation vs. wildtype), RAS mutation status (mutation vs. wildtype), and randomized 1:1 to receive either ramucirumab/TAS102 (arm A) or TAS102 (arm B). Concurrent use of other chemotherapy is not allowed.

Two interim safety analyses will be conducted when 10 and 40 patients are fully documented in arm A after receiving 2 cycles (one 4-week cycle comprises ramucirumab 8mg/kg administered at d1 and d15 and TAS102 35mg/m2 p.o. twice daily administered on d1-5 and d8-12). The analysis will be reviewed by the lead coordinating investigator (Prof. Dr. Kasper) and members of the steering committee and then by the data safety monitoring board. It is not planned to discontinue recruitment for the interim safety analyses.

Arm A (ramucirumab/TAS102) Patients randomized to arm A will receive ramucirumab 8 mg/kg iv over 60 min on d1+15, q4w and TAS102 35mg/m2 p.o. twice daily (BID) d1-5 and 8-12, q4w until progression or intolerance or completion of 6 cycles.

Arm B (TAS102) Patients randomized to arm B will receive TAS102 35mg/m2 p.o. twice daily (BID) d1-5 and 8-12, q4w until progression, intolerance or completion of 6 cycles.

In both arms, tumor assessments (CT or MRI) are performed before enrollment/randomization and then every 8 weeks (every 2nd cycle) during therapy and every 12 weeks during follow-up until progression/relapse, death or end of follow-up. A change from CT into MRI in the follow-up period is possible at any time.

During treatment, clinical visits (blood cell counts, detection of toxicity) will be performed prior to every treatment dose of ramucirumab or every two weeks in arm B or if ramucirumab was discontinued in arm A. Safety of TAS102 +/- ramucirumab will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported. Every 4 weeks during therapy Quality of life (QoL) will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC-QLQ-C30) and the EuroQol 5 dimensions 5-level version (EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic and inoperable, colorectal cancer who has progressed on/after, or did not tolerate, refuse or have contraindications to: fluoropyrimidines, oxaliplatin, irinotecan, anti-angiogenic therapies (bevacizumab, aflibercept, regorafenib or ramucirumab) and if indicated anti-EGFR antibodies (cetuximab or panitumumab).

   Intolerance is defined as a permanent discontinuation of the respective treatment resulting from toxicity
2. Signed informed consent before start of specific protocol procedure
3. Histologically or cytologically documented diagnosis of adenocarcinoma of the colon or rectum
4. Presence of at least one measurable site of disease following RECIST 1.1 criteria
5. ECOG (Eastern Cooperative Oncology Group) performance 0-1
6. Known RAS and BRAF V600E mutational status
7. Life expectancy of at least 3 months
8. Adequate hematological, hepatic and renal function parameters:

   1. Leukocytes ≥3000/mm³, platelets ≥100,000/mm³, neutrophil count (ANC) ≥1500/μL, hemoglobin ≥9 g/dL (5.58 mmol/L)
   2. Adequate coagulation function as defined by International Normalized Ratio (INR) ≤1.5, and a partial thromboplastin time (PTT) ≤5 seconds above the ULN (upper limit of normal) (unless receiving anticoagulation therapy). Patients receiving warfarin/phenprocoumon must be switched to low molecular weight heparin and have achieved a stable coagulation profile prior to first dose of protocol therapy
   3. Serum creatinine ≤1.5 x upper limit of normal or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
   4. Urinary protein ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol)
   5. Bilirubin ≤1.5 x upper limit of normal, AST and ALT ≤3.0 x upper limit of normal, ≤5xULN if liver metastasis present, alkaline phosphatase ≤6 x upper limit of normal
9. Patient able and willing to provide written informed consent and to comply with the study protocol
10. Female and male patients ≥18. Patients in reproductive age must be willing to use adequate contraception during the study and for 7 months after the end of ramucirumab treatment (appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy) or hormonal contraception (implantable, patch, oral). Women who use a hormonal contraception method should use an additional barrier method like IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start (There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.)

Exclusion Criteria:

1. Known hypersensitivity against ramucirumab or TAS102
2. Other known contraindications against ramucirumab, TAS102, or other anti-angiogenic therapies
3. Prior therapy with TAS102
4. Drug-related severe adverse events upon pretreatment with antiangiogenic drugs that would require permanent discontinuation and not allow re-challenge with the same class of drug (i.e. ramucirumab) such as noncontrollable severe hypertension or thromboembolic events
5. Any antineoplastic treatment including irradiation within 14 days (42 days for mitomycin c) prior to start of therapy.
6. Major surgery within 4 weeks of starting therapy within this study, or minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
7. Symptomatic brain metastasis
8. Clinically significant cardiovascular disease

   * NYHA>II°, myocardial infarction within 6 months prior study entry
   * Known clinically significant valvular defect
   * Uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or >100 mmHg diastolic for >4 weeks) despite standard medical management
   * Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy
   * History of deep vein thrombosis (DVT), symptomatic pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy
9. Active clinically serious infections (> grade 2 NCI-CTC version 4.0)
10. Chronic inflammatory bowel disease
11. History of uncontrolled HIV infection or chronic hepatitis B or C
12. Patients with evidence of bleeding diathesis
13. Grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy
14. Receiving chronic antiplatelet therapy, including aspirin (once daily aspirin use (maximum dose 325 mg/day) is permitted), nonsteroidal anti-inflammatory drugs (including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents
15. History of gastrointestinal perforation or fistulae in past 6 months or risk factors for perforation
16. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy
17. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix or bladder, or low/intermediate risk prostate cancer (Gleason score ≤7) with normal PSA levels
18. Any condition that could jeopardize the safety of the patient and their compliance of the study
19. Medical, psychological or social conditions that may interfere with the participation in the study
20. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or ascites.

    Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
21. On-treatment participation in another clinical study or received investigational drug therapy in the period 30 days prior to inclusion and during the study
22. Subject pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment
23. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
24. Any other concurrent antineoplastic treatment including irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 4 years
  Overall survival according to Kaplan-Meier

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  ORR defined as the proportion of patients with complete or partial remission according to RECIST 1.1
Disease control rate (DCR) | Up to 4 years
  DCR defined as the proportion of patients with complete or partial remission and stable disease according to RECIST 1.1
Progression-free survival (PFS) | Up to 4 years
  PFS, defined as the time from enrollment/randomization to the first occurrence of progression, as determined by the investigator using CT criteria, or death from any cause
Overall survival (OS) rate at different time points | 6 months and 1 year
  OS rate at 6 and 12 months, defined as patients who are alive after at 6 and 12 months, respectively
Efficacy (ORR) subgroup | Up to 4 years
  Efficacy (ORR) in patients who develop neutropenia grade ≥2 (ANC ≤1500/μl) in cycle 1
Efficacy (PFS) subgroup | Up to 4 years
  Efficacy (PFS) in patients who develop neutropenia grade ≥2 (ANC ≤1500/μl) in cycle 1
Efficacy (OS) subgroup | Up to 4 years
  Efficacy (OS) in patients who develop neutropenia grade ≥2 (ANC ≤1500/μl) in cycle 1
Quality of life I (QoL) | Up to 1 year
  Quality of life (QoL) as measured by EORTC-QLQ-C30 at d1 of each cycle and on EOT (end of treatment).
Quality of life II (QoL) | Up to 1 year
  Quality of life (QoL) as measured by EQ-5D-5L at d1 of each cycle and on EOT.

OTHER OUTCOMES:
Explorative: Overall response rate (ORR) | Up to 4 years
  ORR according to gene expression, mutational profiles, plasma biomarkers and radiologic analysis
Explorative: Overall survival (OS) | Up to 4 years
  OS according to gene expression, mutational profiles, plasma biomarkers and radiologic analysis
Explorative: Progression-free survival (PFS) | Up to 4 years
  PFS according to gene expression, mutational profiles, plasma biomarkers and radiologic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (28):
- Germany (28):
  - MVZ Gesundheitszentrum St. Marien GmbH, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charité - Universitätsmedizin Berlin Campus Mitte, Berlin
  - MVZ Seestrasse, Berlin
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Hamburg Barmbek, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Marien Hospital Herne, Herne
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg
  - Tagestherapiezentrum am ITM Universitätsmedizin Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universität München-Großhadern, München
  - Unversitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - MedCenter Nordsachsen, Schkeuditz
  - Leopoldina Krankenhaus, Schweinfurt
  - MVZ Klinik Dr. Hancken GmbH, Stade
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Wilhelmshaven, Wilhelmshaven
  - Hämatologisch-Onkologische Praxis, Würselen

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared